CLINICAL TRIAL: NCT00196638
Title: Multicentric Trial Comparing Three Therapeutical Strategies in Patients With Acute Primary HIV Infection.ANRS 112 INTERPRIM
Brief Title: Multicentric Trial Comparing Three Therapeutical Strategies in Patients With Acute Primary HIV Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 112 INTERPRIM
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections; Primary Acute Infection
Keywords: HIV infections; Primary acute infection; Interferon-alpha
MeSH Terms: conditions — HIV Infections | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Antiretroviral combination (drugs)
Drug: Pegylated Interferon alpha (drug)

SUMMARY:
Treatment of acute primary HIV infection may improve long-term outcome. However, optimal treatment is still debated. The ANRS 112-INTERPRIM trial evaluates three different therapeutical strategies, combining permanent or intermittent HAART and a cytokine, interferon alpha, in order to determine which combination allows the best control of HIV viremia after 24 weeks of antiretroviral treatment interruption

DETAILED DESCRIPTION:
Treatment of acute primary HIV infection may improve long-term outcome. However, optimal treatment is still debated. The main objective of this multicentric randomized phase II/III study is to compare HIV viremia 92 and 96 weeks after acute primary HIV infection, between patients treated with 3 different strategies. In the first group, patients receive antiretroviral drugs (HAART) continuously up to week 72. In the second group, patients receive HAART continuously up to week 36, then intermittently up to week 72. In the third group, patients receive HAART as in group II, and pegylated interferon alpha is administered for the initial 14 weeks, then for 3 weeks at each of the 3 HAART interruption between week 36 and week 72. All patients are monitored without any HAART up to week 96. Enrolled patients have circulating p24 antigen and/or HIV viremia, an uncompleted HIV western blot, between 18 and 65 years old, and agree to participate to the study. They should have received no antiretroviral drugs, not be pregnant, without neuro-psychological or autoimmune disorders, without chronic hepatitis. Secondary objectives of the study are: the quality of immune restoration, the anti-HIV immune response, safety and adhesion to treatment. A total of 90 patients (30 in each group) have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* P24 antigen with positive neutralization or positive plasma HIV RNA
* Negative or not complete Western Blot
* With symptoms or not
* Written informed consent

Exclusion Criteria:

* Previous antiretroviral treatment
* Pregnancy
* Biological abnormalities
* Hepatitis C or B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-05; Study Completion 2006-03

PRIMARY OUTCOMES:
Plasma HIV RNA at Week 92 and 96 (mean)

SECONDARY OUTCOMES:
Plasma HIV RNA kinetics after treatment interruption
CD4 cell count
Proviral DNA
Adherence

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Emilie, MD, Principal Investigator — Hôpital Antoine Béclère, Clamart, France; Genevieve Chene, MD, PhD, Study Director — INSERM U593, Bordeaux, France.